CLINICAL TRIAL: NCT02626481
Title: A Multicenter Open Label Phase II Study of Daratumumab in Combination With Dexamethasone in Multiple Myeloma Resistant or Refractory to Bortezomib and Lenalidomide and Pomalidomide - an IFM 2014-04 Study
Brief Title: Study of Daratumumab in Combination With Dexamethasone in Resistant or Refractory Multiple Myeloma
Acronym: IFM2014-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Janssen, LP (Industry); Intergroupe Francophone du Myelome (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015_29; 2015-002221-19 (EudraCT Number)
Record Dates: First submitted 2015-11-16; First posted 2015-12-10 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Cancer; refractory; daratumumab
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — daratumumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daratumumab + Dexamethasone (Experimental): patients treated with Daratumumab (16 mg/kg) and Dexamethasone (40 or 20 mg regarding age of patient)
  Interventions: Drug: Daratumumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — patients treated with Daratumumab (16 mg/kg) and Dexamethasone (40 or 20 mg regarding age of patient)
  Other Names: Experimental Arm
Drug: Dexamethasone — patients treated with Dexamethasone (40 or 20 mg regarding age of patient)
  Other Names: Experimental Arm

SUMMARY:
This study is a Multicentre, Open-label, Phase II study of Daratumumab and Dexamethasone in MM patients. Eligible patients must have a symptomatic RRMM with a measurable disease, resistant or refractory to Bortezomib and Lenalidomide and Pomalidomide.

There is no dose escalation phase, as the MAxiamal Tolerated Dose (MTD) and drug scheduling have already been determined in previous phase 1-2 dose escalation studies. There is no randomization.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is the second most common haematological malignancy (after non-Hodgkin's lymphoma), representing 1% of all cancers and 2% of all cancer deaths. Despite the increased efficacy of first-line agents, the majority of patients will eventually relapse and become resistant to all classes of available therapies. With over 15,000 deaths from MM expected in 2014 in the United states of America (USA) alone, there remains a need for novel therapies for the treatment of refractory MM that can improve outcome Daratumumab is an IgG1ĸ human mAb that specifically recognizes the CD38 epitope. Daratumumab binds to the C-terminus of CD38. It is produced in a recombinant Chinese Hamster Ovary (CHO) cell line. Standard mammalian cell culture and purification technologies are employed in the manufacture of Daratumumab. Daratumumab targets directly the tumour cells by selectively binding to CD38 receptors, present in high levels on malignant plasma cells in multiple myeloma. While binding of Daratumumab antibody to CD38 in vitro has some effect on enzyme activity (inhibiting cyclase and stimulating hydrolase activity), the main effect of Daratumumab antibody binding to CD38+ myeloma cell lines is lysis and cell death through complement dependent cytotoxicity (CDC), through antibody dependent cell-mediated cytotoxicity (ADCC) or antibody-dependent cell phagocytosis (ADCP), or by direct apoptosis following crosslinking of the antibody molecules. These mechanisms are likely to be involved in Daratumumab activity in vivo, although the primary mechanism of action in patients is not fully elucidated. Importantly, Daratumumab-induced ADCC and CDC was not affected by the presence of bone marrow stromal cells, indicating that Daratumumab can effectively kill MM tumour cells in a tumour-preserving bone marrow microenvironment. In vivo, Daratumumab was highly active and interrupted xenograft tumour growth at low dosing. Daratumumab has demonstrated activity in myeloma as a single agent in small phase I/II studies and in combination with Lenalidomide and Dexamethasone where it enhanced the potency of other MM drugs such as Lenalidomide offering an interesting alternative to chemotherapy in myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and voluntarily sign an informed consent form
2. Must be able to adhere to the study visit schedule and other protocol requirements
3. Age ≥18 years
4. Life expectancy > 6 months
5. Patients must have relapsed myeloma, and previously treated with Bortezomib, Lenalidomide, and Pomalidomide treatment, and being resistant or refractory to Bortezomib and Lenalidomide and Pomalidomide treatment, defined as follows:

   5.1. Any number of prior therapies 5.2. Patients must have Progressive Disease as defined by the IMWG as one of the following (Kyle, 2009):

   Increase of 25% from lowest response value in any one or more of the following:
   * Serum M-component (absolute increase must be ≥ 0.5 g/100 ml)b and/or Urine M-component (absolute increase must be ≥ 200 mg per 24 h) and/or
   * Only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved
   * FLC levels (absolute increase must be > 10 mg/l). Bone marrow plasma cell percentage (absolute % must be ≥ 10%)
   * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
   * Development of hypercalcemia (corrected serum calcium > 11.5 mg/100 ml) that can be attributed solely to the plasma cell proliferative disorder 5.3. Patients must have undergone prior treatment with Bortezomib and Lenalidomide and Pomalidomide:
   * They must have received at least two cycles of therapy
   * Either at diagnosis or relapse
   * Either in separate regimens or within the same regimen
   * The line of treatment with Bortezomib and/or Lenalidomide and/or Pomalidomide does not need to be the very last line of prior therapy
6. Patients must have a clearly detectable and quantifiable monoclonal M-component value:

   IgG (serum M-component > 10g/l) IgA (serum M-component >5g/l) IgD (serum M-component > 0.5g/l) Light chain (serum M-component >1g/l or Bence Jones > 200mg/24H) In patients without measurable serum and urine M-protein levels when the absolute serum FreeLight chain (sFLC) is ≥100 mg/l and an abnormal sFLC K/λ ratio (<0.26 and >1.65) is found (Dispenzieri, 2008).
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
8. Adequate bone marrow function within 5 days prior to 1st drug intake (cycle1, day 1, C1D1), without transfusion nor growth factor support within 5 days prior to 1st drug intake , defined as:

   Absolute neutrophils ≥ 1000/mm3 Platelets ≥ 50000/mm3 Haemoglobin ≥ 8.5g/dl
9. Adequate organ function defined as:

   Serum creatinine clearance (Cockcroft-Gault formula) ≥30 ml/min Serum SGOT or SGPT < 3.0 X upper limit of normal (ULN) Serum total bilirubin < 2.0 mg/dL
10. Wash out period of at least 2 weeks from previous antitumor therapy or any investigational treatment or 5 half-lives from previous antibodies.
11. Women who are partners of men and of childbearing potential must be practicing one of the following methods of birth control: subcutaneous hormonal implant, levonorgestrel releasing intra-uterine system, medroxyprogesterone acetate depot, tubal sterilization, ovulation inhibitory progesterone only pills, or sexual intercourse with a vasectomized male partner (vasectomy must be confirmed by 2 negative semen analyses). Or women will commit to absolute and continuous abstinence confirmed to her physician on a monthly basis. Childbearing potential*. Contraception will start during therapy including dose interruptions, for 4 months after discontinuation of Daratumumab.

    * Criteria for women of childbearing potential :

This protocol defines a female of childbearing potential as a sexually mature woman who:

1. has not undergone a hysterectomy or bilateral oophorectomy or
2. has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months) 12. A woman of childbearing potential must have 2 negative serum or urine pregnancy tests at Screening, first within 28 days prior to dosing and the second within 48 hours prior to dosing, and remain on a highly effective method of birth control. The two methods of reliable contraception must include one highly effective method and one additional effective (barrier) method. FCBP must be referred to a qualified provider of contraceptive methods if needed. The following are examples of highly effective and additional effective methods of contraception:

   * Highly effective methods:

     * Intrauterine device (IUD)
     * Hormonal (birth control pills, injections, implants)
     * Tubal ligation
     * Partner's vasectomy
   * Additional effective methods:

     * Male condom
     * Diaphragm
     * Cervical Cap 13. Serum (urine in the case where serum is not possible in a timely manner) pregnancy test to be performed for all women of childbearing potential regularly during the study,. In addition, a pregnancy test may be done at any time during the study at the discretion of the investigator if a subject misses a period or has unusual menstrual bleeding.

       14. A woman of childbearing potential must remain on a highly effective method of birth control. Contraception must begin 4 weeks before initiating treatment with Daratumumab, during therapy, during dose interruptions and continuing for 4 months following discontinuation of Daratumumab. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy.

       15. A man who has not had a vasectomy and who is sexually active with a woman of childbearing potential must agree to use a barrier method of birth control eg, condom with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study, for 4 months following discontinuation of Daratumumab. The exception to this restriction is that if the subject's female partner is surgically sterile, a second method of birth control is not required.

       16. Subjects affiliated with an appropriate social security system.

Exclusion Criteria:

1. Target disease exceptions:

   * Solitary bone/solitary extramedullary plasmocytoma
   * Patients with non-secretory MM and non-measurable MM
   * Evidence of central nervous system (CNS) involvement
2. Medical history and Concurrent disease:

   o Subjects with prior (≤ 5 years) or concurrent invasive malignancies except the following: Adequately treated basal cell or squamous cell skin cancer Incidental finding of low grade (Gleason 3+3 or less) prostate cancer Any cancer from which the subject has been disease free for at least 3 years.
   * Subject with known/underlying medical conditions that, in the investigator's opinion would make the administration of the study drug hazardous (ie: uncontrolled diabetes or uncontrolled coronary artery disease)
   * Any uncontrolled or severe cardiovascular or pulmonary disease determined by the investigator including:

   NYHA functional classification III or IV congestive heart failure LVEF ( Left Ventricular Ejection Fraction) ≥45% Uncontrolled angina, hypertension or arrhythmia Myocardial infarction in the past 6 months
   * Subjects with grade 2 or greater peripheral neuropathy (as per NCI-CTCAEv4.0)
   * Subject is a woman who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 4 months after the last dose of any component of the treatment regimen. Or, subject is a man who plans to father a child while enrolled in this study or within 4 months after the last dose of any component of the treatment regimen.
   * Known positive for HIV or active hepatitis B or C.
   * Subjects with psychiatric illnesses or social situations that would preclude them understanding the informed consent, study compliance or the ability to tolerate study procedures and/or study therapy
   * Subjects with known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for patients suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.
   * Subjects with a history of moderate or severe persistent asthma within the past 2 years (see appendix), or with uncontrolled asthma of any classification at the time of screening (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study).
3. Physical and laboratory test findings:

   * Patients on dialysis or with a Creatinine clearance < 30mL/min
   * SGOT or SGPT >3ULN
4. Prohibited prior therapies

   * Prior local irradiation within two weeks before first dose
   * Previous anti-CD38 therapy.
5. Allergies and Adverse Drug Reaction:

   o Hypersensitivity to Dexamethasone that would prohibit treatment with study therapy
6. Refusal to consent or protected by a legal regime (guardianship, trusteeship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-12-28 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Number of best Overall Response using the IMWG response criteria | 60 months
  best Overall Response Rate (ORR, PR or better) using the IMWG response criteria.

SECONDARY OUTCOMES:
Number of patients with treatment-related adverse events as assessed by CTCAE v4.0 | 60 months
  Assess safety by type, frequency, severity, relationship of adverse events to study treatment and changes in vital signs, physical exams. Incidence of Treatment Emergent Adverse Event (TEAE), Serious Adverse Event (SAE) and laboratory abnormalities using National Cancer Institute (NCI) common toxicity criteria (CCTAE V4).
Number of patients who reach Very Good Partial Response and Complete using IMWG response criteria | 60 months
  Response rate (VGPR and CR) to Daratumumab and Dexamethasone in the study population using IMWG response criteria.
Rate of Overall Survival (OS) | 60 months
  Determine the OS (from the date of inclusion to last date of follow-up) of patients treated with Daratumumab+ Dexamethasone.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Facon, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (41):
- Belgium (4):
  - AZ ST Jan hematology department, Bruges
  - Hematologie Laarbeeklaan, Brussels
  - Jules Bordet Institute, Brussels
  - CHU Dinant Godinne | UCL Namur asbl, Yvoir
- France (37):
  - CHRU - Hôpital du Bocage (Amiens), Amiens
  - CHRU-Hôpital Sud d'Amiens, Amiens
  - Hôpital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hôpital du Haut Lévêque Centre François Magendie, Bordeaux
  - Clinique - ICH CHU de Brest Hôpital Morvan, Brest
  - CHRU Côte de Nacre, Caen
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Hôpital d'instruction des armées Percy, Clamart
  - Hématologie Clinique CHU DIJON, Dijon
  - Centre Hospitalier Général, Dunkirk
  - CHRU, Hôpital A.Michallon, Grenoble
  - Médecine interne Centre hospitalier départemental, La Roche-sur-Yon
  - Service d'Hématologie CHV André Mignot, Le Chesnay
  - CHRU , Hôpital Claude Huriez, Lille
  - Sce Hématologie Thérapie Cellulaire CHU Limoges, Limoges
  - Institut Paoli Calmette, Marseille
  - Hopital J Monod Sce Rhumato Nord, Montivilliers
  - Service Hématologie CHRU Montpellier, Montpellier
  - Hopital E Muller, Mulhouse
  - Maladies du sang CHRU Hôtel Dieu, Nantes
  - URC/CIC Paris Descartes Necker-Cochin, Paris
  - Curie Institut, Paris
  - Hôpital Saint-Louis, Paris
  - CHU - Hôpital St Antoine, Paris
  - Unité de Recherche Clinique - CH Périgueux, Périgueux
  - Centre Hospitalier Lyon sud, Pierre-Bénite
  - CHU de la milétrie, Poitiers
  - Hôpital R.Debré, Reims
  - Hôpital de Pontchaillou, Rennes
  - Service Hématologie Centre Hospitalier Yves le Foll, Saint-Brieuc
  - Service d'Hématologie Clinique Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Département d'Hématologie et Oncologie Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hématologie CHRU IUCT Oncopole, Toulouse
  - Onco-hématologie CHRU Hôpital Bretonneau, Tours
  - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - service hématologie CH Bretagne Atlantique, Vannes